CLINICAL TRIAL: NCT07153393
Title: A Single-Arm Study of HTIC (Heterologous Type I Collagen) Intradermal Injections for the Medical Treatment of Dermal Defects Due to Scarring, Hypotonia, and Hypotrophy
Brief Title: A Clinical Study Testing How Well the Medical Device HTIC (a Type of Animal-derived Collagen) Works in Treating Skin Problems, Such as Scars, Loss of Firmness, and Volume in Certain Areas of the Face and Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Studi Dermatologici S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTIC-10-22
Record Dates: First submitted 2025-08-22; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Skin Aging of Face and Hands; Cicatrix; Scars; Atrophic Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HTIC - Adults 18-50, Fitzpatrick I-V, Mild to Moderate Skin Volume Loss (Experimental): In this arm, 45 subjects of both sexes, aged between 18 and 50 years, of Caucasian ethnicity with Fitzpatrick skin phototype ranging from I to V, will receive treatment with the experimental medical device HTIC. Participants will be selected based on the presence of skin defects characterized by mild to moderate volume loss due to acne scars, other skin lesions, or photoaging. Inclusion requires a minimum score of 2 according to the Modified Fitzpatrick Wrinkle Scale. The treatment involves subcutaneous administration of HTIC, consisting of injecting 0.1 ml per intradermal site at intervals of approximately 2 cm.
  Interventions: Device: Type I Bovine Collagen (HTIC)

INTERVENTIONS:
Device: Type I Bovine Collagen (HTIC) — HTIC is a sterile collagen powder (100 mg) contained in a glass vial, which is diluted by adding 5 ml of saline solution (0.9% sodium chloride solution) to obtain a suspension. This suspension will be prepared immediately before treatment. The procedure consists of performing a few microinjections of the product (0.1 ml per injection) into the dermis at intervals of approximately 2 cm, using a very fine needle (30G/32G, 4 mm) in the areas to be treated (face, neck, décolleté, and hands).

SUMMARY:
This clinical trial aims to evaluate the efficacy of the experimental medical device HTIC, which contains Type I collagen of animal origin, in treating skin defects such as scars, loss of tone, and volume in certain areas of the face and body. HTIC is administered through an injection technique applied under the skin. The main research question is: "Is it possible to achieve clinical improvement of skin defects through the use of the experimental device HTIC?"

Additionally, the study has the following secondary objectives:

* To assess any discomfort experienced during administration;
* To evaluate the subject's level of satisfaction following the entire treatment;
* To assess the safety and tolerability of the experimental device HTIC. HTIC is a sterile powder composed solely of animal-derived collagen (heterologous bovine Type I collagen, allergen-free and compliant with current regulations), packaged in 10 ml glass vials. Each vial contains 100 mg of sterile bovine Type I collagen powder.

The trial will be conducted at a single site in Italy, specifically at the Federico II University Hospital. A total of 45 subjects will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (age between 18-50 years).
2. Subjects in good health.
3. Subjects that presented skin atrophy from acne scarring, other injury, or photo-aging (from mild to moderate).
4. Subjects with a score at least 2 according to the Modified Fitzpatrick Wrinkle Scale (MFWS).
5. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Ethics Committee (EC).

Exclusion Criteria:

Subjects will not be enrolled in the study if any of the exclusion criteria listed below are met:

1. Pregnant or breastfeeding.
2. Subjects that had undergone other medical invasive aesthetic treatments for the last 18 months before the enrolment.
3. Subjects with acne.
4. Subjects with seborrheic skin.
5. Subjects with normotonic, normoelastic, and normotrophic skin.
6. Subjects with autoimmune connective tissue disorders (connectivopathies).
7. Subjects with a tendency to develop hypertrophic or keloid scars.
8. Subjects undergoing immunosuppressive therapy.
9. Any cutaneous pathology of infectious, inflammatory, viral and vascular type affecting the treated area.
10. History of allergy or hypersensitivity to any component of the study devices.
11. Performing permanent filler in the past.
12. Use of any therapeutic agent for photoaging or skin rejuvenation within 15 days from the enrolment.
13. Smoking.
14. Wound healing disorders.
15. Participation in other clinical studies.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Measurement of the global aesthetic change between Visit 0 (Screening and Baseline) and Visit 5 (7 days) after the last HTIC injection | Screening and Baseline visit (day 0) and Visit 5 ( 7 days after the last HTIC injection_Visit 4)
  The aesthetic change will be assessed by the Investigator using a 5-point Global Aesthetic Improvement Scale (GAIS) by comparing the subject's photograph taken prior and after the treatment.
  (Scale values: from 1 to 5.) Lower scores indicate a better outcome (greater aesthetic improvement), while higher scores indicate a worse outcome (no improvement or worsening).

SECONDARY OUTCOMES:
Clinical skin assessment together with photographic evaluation at Visit 0 and Visit 5, using the 7-point Modified Fitzpatrick Wrinkle Scale (MFWS). | Screening and Baseline visit (day 0) and visit 5 (7 days after the last HTIC injection_V4)
  Modified Fitzpatrick Wrinkle Scale (MFWS) Scale values: from 0 to 3 Lower scores indicate a better aesthetic outcome (fewer or less severe wrinkles), while higher scores reflect a worse outcome (more prominent or deeper wrinkles).
Self-assessment of the subject's satisfaction with the procedure using a Visual Analog Scale (VAS), ranging from 0 (very satisfied) to 10 (very dissatisfied), at Visit 5 compared to Visit 1 | Visit 5 (7 days from the last HTIC injection) and Visit 1(≤7 days from Screening & baseline visit_day 0)
  Visual Analog Scale (VAS) Scale range: 0 to 10, 0 (very satisfied) and 10 (very dissatisfied)
Self-assessment of pain by the subject during the injection treatment at Visits 1, 2, 3, and 4, using a Visual Analog Scale (VAS) after each treatment | At visit 1(≤7 days from Screening & Baseline visit_day 0), Visit 2 (7 days from V1), Visit 3(7 days from V2) and Visit 4 (7 days from V3)
Collection and evaluation of the rate of related adverse events (AEs) occurring during the study. | at Screening & Baseline visit (day 0), Visit 1(≤7 days from V0), Visit 2 (7 days from V1), Visit 3 (7 days from V2), Visit 4 (7 days from V3) and Visit 5 (7 days from V4_the last HTIC injection)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Federico II, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No